CLINICAL TRIAL: NCT06955819
Title: GUTPROH Trial: A Double-Blind, Randomized, Placebo-Controlled Study of Probiotic-Multiherb Formula for Self-Reported Constipation Symptoms in Community-Dwelling Adults
Brief Title: GUTPROH: Probiotic-Herbal Formula for Self-Reported Constipation in Community Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Collaborators: Chinese Aging Well Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025BJYYEC-KY016-02
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-03

CONDITIONS: Functional Constipation (FC)
Keywords: Probiotic; Herbal powder; Functional constipation; Gut microbiota; Randomized controlled trial; Placebo control; Community population; Efficacy evaluation; Mechanism exploration
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo Control Group (Placebo Comparator): Participants in the placebo control group will take a blank matrix powder. The dosage and administration method are the same as those of the experimental groups. That is, they will take a certain amount of the powder twice a day (the same frequency as the probiotic powder intake in the experimental groups) and once every other day (the same frequency as the herbal powder intake in the experimental groups). The blank matrix powder does not contain probiotics or herbal powder but is designed to have the same appearance as the experimental products. This is to eliminate the placebo effect and serve as a baseline for comparison. During the 12 - week study period, participants in this group also need to record their daily defecation, diet, and adverse reactions, and undergo the same fecal gut microbiota examination and serum mass spectrometry non - targeted metabolomics measurement at week 0, week 4, and week 12 as the experimental groups.
  Interventions: Other: Placebo Intervention
- Probiotic Intervention Group (Experimental): Subjects in this group will consume Zhigu Zhijian (QingzhiningTM) probiotic powder. The dosage is 2g per time, and it should be taken twice a day, specifically after breakfast and dinner. The probiotic powder is taken with lukewarm water (water temperature ≤ 30℃). The purpose of this intervention is to explore the individual effect of the probiotic on improving defecation and gut microbiota in participants with a need for better bowel movements. The intervention period is 12 weeks. Similar to the other groups, participants are required to keep daily records of defecation - related information, diet, and adverse reactions. They also need to participate in the same series of examinations at week 0, week 4, and week 12 to assess the impact on gut microbiota and metabolic function.
  Interventions: Dietary Supplement: Probiotic Intervention
- Probiotic with Herbal Powder Intervention Group (Experimental): Participants in this group will take Zhigu Zhijian (QingzhiningTM) probiotic powder at a dosage of 2g per time, twice a day (after breakfast and dinner), and Zhigu Zhijian (QingzhiningTM) herbal powder at a dosage of 15g per time, once every other day (before breakfast). The probiotic powder should be taken with lukewarm water (water temperature ≤ 30℃), and the herbal powder should be taken after being brewed with boiling water. This intervention aims to evaluate the combined effect of the compound probiotic and herbal powder on improving defecation problems and gut microbiota in subjects with defecation - related demands. The duration of the intervention is 12 weeks. During this period, participants need to record their daily defecation frequency, defecation status, fecal characteristics, daily diet, and report any adverse reactions. They also need to participate in the same series of examinations at week 0, week 4, and week 12.
  Interventions: Dietary Supplement: Probiotic with Herbal Powder Intervention

INTERVENTIONS:
Other: Placebo Intervention — Subjects will be given a blank matrix powder with the same appearance as the products in the experimental groups, which does not contain probiotics or herbal powder. The dosage, frequency, and administration method are exactly the same as those in Experimental Group. Intervention duration will be 12 weeks, carried out synchronously with the experimental groups to ensure the consistency of research conditions.
  Arms: Placebo Control Group
Dietary Supplement: Probiotic Intervention — Subjects will take Zhigu Zhijian (QingzhiningTM) probiotic powder, 2g per sachet, twice a day, one sachet after breakfast and one after dinner, taken with lukewarm water (water temperature ≤ 30℃). Intervention duration will also be 12 weeks, for parallel comparison with other groups.
  Arms: Probiotic Intervention Group
Dietary Supplement: Probiotic with Herbal Powder Intervention — Subjects in this group will be given Zhigu Zhijian (QingzhiningTM) probiotic powder and Zhigu Zhijian (QingzhiningTM) herbal powder. The probiotic powder is 2g per sachet, taken twice a day, one sachet after breakfast and one after dinner, and should be taken with lukewarm water (water temperature ≤ 30℃). The herbal powder is 15g per sachet, taken once every other day before breakfast, and should be taken after being brewed with boiling water. Intervention duration will be last for 12 weeks to ensure sufficient time to observe the long - term effects on defecation and gut microbiota.
  Arms: Probiotic with Herbal Powder Intervention Group

SUMMARY:
The goal of this clinical trial is to evaluate the effects of probiotic combined with or without herbal powder on relieving constipation and improving the gut microbiota in community - dwelling people with a demand for improved bowel movements through human feeding trials, and to explore their potential mechanisms of action.

The main research questions are as follows:

Can the probiotic combined with or without herbal powder significantly increase the frequency of defecation in subjects, and at the same time improve fecal characteristics and defecation conditions? Can the the probiotic combined with or without herbal powder regulate the gut microbiota? What are the biological mechanisms by which the probiotic combined with or without herbal powder improve constipation and gut microbiota function? Researchers will compare experimental group 1 (taking the compound probiotic combined with herbal powder), experimental group 2 (taking probiotics alone) with the placebo control group (taking an identical - looking blank matrix powder) to observe their effects on defecation and the gut microbiota.

The main tasks for participants include:

Taking the compound probiotic combined with herbal powder (experimental group 1), probiotics alone (experimental group 2), or blank matrix powder (placebo control group) as required for 12 weeks.

Recording daily defecation frequency, defecation conditions, fecal characteristics, and daily diet, and reporting any adverse reactions.

Longitudinal monitoring employs serial assessments comprising: 1) physical examinations (mental status/vital signs); 2) laboratory diagnostics (hematology/urinalysis/fecal routine tests, hepatic-renal-metabolic panels); 3) ECG and abdominal ultrasonography; and 4) advanced analyses (gut microbiome sequencing and serum metabolomic profiling via LC/MS/MS).

ELIGIBILITY:
Inclusion Criteria:

* Aged 35 years or older.
* Self - reported good comprehensive physical health status. Have complaints of irregular bowel movement frequency and a need for improved defecation, or have a spontaneous defecation frequency of less than 3 times per week in the 2 weeks before administration, or meet two or more of the following Rome IV criteria for functional constipation (FC): ① >25% of defecations are difficult; ② >25% of defecations are dry, hard, or pellet - shaped; ③ >25% of defecations have a sense of incomplete evacuation; ④ >25% of defecations have a feeling of anorectal obstruction or blockage; ⑤ >25% of defecations require manual assistance; ⑥ Fewer than 3 spontaneous defecations per week.
* Provide written informed consent voluntarily before the study and be able to fill out the subject log card and research questionnaire as required by the trial protocol.

Exclusion Criteria:

* Frail elderly people with a score of ≥3 on the FRAIL Frailty Screening Scale.
* Self - reported presence of loose stools.
* Those who have undergone surgery within 30 days, had an acute gastrointestinal disease within 30 days, or have been diagnosed with severe organic diseases causing defecation difficulties (such as colon cancer, intestinal obstruction, inflammatory bowel disease, etc.).
* Patients with severe systemic diseases in the acute phase of cardiovascular, liver, kidney, and hematopoietic systems.
* Patients with symptoms of yin deficiency and internal heat, such as dry mouth, night sweats, restlessness of the five centers (palms, soles, and chest), hard and dry stools with bad breath, red tongue with yellow coating.
* Those who have taken antibiotics within 30 days before the start of the trial.
* Those who have taken probiotics, fermented products, other laxative drugs, or health supplements within 14 days before the start of the trial (i.e., during the wash - out period).
* Those who have not signed the informed consent form. Other situations considered unsuitable for enrollment by the researchers.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in spontaneous defecation frequency | From the start of intervention (week 0) to the end of the 12 - week intervention period.
  The number of spontaneous bowel movements per week. An increase in the frequency of spontaneous defecation in the experimental groups compared to the placebo control group would indicate a potential positive effect of the interventions.

SECONDARY OUTCOMES:
Improvement in fecal characteristics | From the start of intervention (week 0) to the end of the 12 - week intervention period.
  Evaluated using the Bristol Stool Form Scale (a 1-to-7 scale, where 1 represents the most abnormal stool form [e.g., separate hard lumps] and 7 represents the most watery/diarrheal form). An improvement in fecal characteristics is defined as moving from lower-scored forms (1-2, indicating constipation-predominant states) to higher-scored, more "normal" forms (3-5, indicating optimal bowel movement consistency). Higher scores within this context (toward the 3-5 range) signify a better outcome, suggesting a beneficial impact on defecation.
Alteration in defecation status | From the start of intervention (week 0) to the end of the 12 - week intervention period.
  Assessed using a defecation difficulty scoring system (a 0-to-3 scale, where 0 indicates no defecation difficulty and 3 indicates severe defecation difficulty). The scale includes the following scores: 0 = no difficulty; 1 = mild difficulty (e.g., occasional straining); 2 = moderate difficulty (e.g., frequent straining or incomplete evacuation); 3 = severe difficulty (e.g., prolonged straining, use of laxatives, or inability to defecate without assistance). In this scoring system, higher scores represent worse outcomes (i.e., greater defecation difficulty), whereas a reduction in the score (e.g., from 3 to 1) indicates an improvement in defecation status.

OTHER OUTCOMES:
Changes in Gut Microbiota | The start of the intervention (week 0), week 4 and week 12 of the intervention.
  Analyze the changes in the quantity and proportion of bacterial genera such as Bifidobacterium, Lactobacillus, Clostridium perfringens, Enterobacter, Enterococcus, and Bacteroides through 16s sequencing of feces, to evaluate the regulatory effects of the compound probiotic combined with herbal powder and probiotics alone on the gut microbiota. From the start of the intervention (week 0) to week 4 and week 12 of the intervention.
Changes in Gut Microbiota Metabolic Remodeling Indicators | The start of the intervention (week 0), week 4 and week 12 of the intervention.
  Use serum mass spectrometry non - targeted metabolomics to detect changes in the metabolites of the gut microbiota, comprehensively determine whether the metabolic function of the gut microbiota has been improved, and explore the time - series change rules at week 4 and week 12. From the start of the intervention (week 0) to week 4 and week 12 of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Sun, Ph.D, Principal Investigator — Beijing Hospital